CLINICAL TRIAL: NCT07353411
Title: A Prospective, Single-center, Single-arm Clinical Study to Evaluate the Effectiveness and Safety of Single-port Robotic-assisted Subcutaneous Gland Resection in Males
Brief Title: To Evaluate the Effectiveness and Safety of Single-port Robotic-assisted Subcutaneous Gland Resection in Males
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DQ-GYN-Robot-20251010
Record Dates: First submitted 2025-12-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Gynecomastia
Keywords: Single-port Robotic-assisted subcutaneous gland resection
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Intervention Model Description: Single-port Robotic-assisted Subcutaneous Gland Resection for males in the treatment of gynecomastia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the single-port robotic-assisted subcutaneous gland resection group (Experimental): the single-port robotic-assisted subcutaneous gland resection in the management of gynecomastia
  Interventions: Procedure: Single-port Robotic-assisted Subcutaneous Gland Resection in males

INTERVENTIONS:
Procedure: Single-port Robotic-assisted Subcutaneous Gland Resection in males — Single-port Robotic-assisted Subcutaneous Gland Resection for males in the treatment of gynecomastia.

SUMMARY:
The new technology of robotic surgery system, as an emerging technology, has shown certain application prospects in breast surgery. However, the new technology of robotic surgery system in China in the treatment of gynecomastia is still in the exploratory stage and needs to be further improved. This prospective, single-center, single-arm clinical study was conducted to use the single-port robot and evaluate the effectiveness and safety of the subcutaneous gland resection in the treatment of gynecomastia.

DETAILED DESCRIPTION:
The new technology of robotic surgery system, as an emerging technology, has shown certain application prospects in breast surgery. However, the new technology of robotic surgery system in China in the treatment of gynecomastia is still in the exploratory stage and needs to be further improved. This prospective, single-center, single-arm clinical study was conducted to use the single-port robot and evaluate the effectiveness and safety of the subcutaneous gland resection in the treatment of gynecomastia.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients, aged 18-75 years old;
2. Preoperative breast ultrasound indicates male breast development, and breast enlargement symptoms persist for more than 1 year;
3. Primary male breast development that has been unresponsive to drug treatment, or those who refuse drug treatment;
4. According to Gynecomastia's surgical indications, refer to the "2023 Expert consensus on the clinicaldiagnosis and treatment of gynecomastia in China" Simon grading of male breast development IIb or above;
5. Due to social pressure or severe psychological burden caused by symptoms such as breast pain, those who have a strong desire for surgery may experience psychological burden caused by the disease and actively request surgery;
6. Individuals without serious accompanying diseases;
7. Suspected malignant transformation;
8. No other serious underlying diseases in the past;
9. The surgical procedure includes a single hole robot (intraperitoneal endoscopic single hole surgical system SP1000) for subcutaneous gland resection of the breast;
10. Participants are able to understand the research process, voluntarily join the study, sign informed consent forms, have good compliance, and cooperate with follow-up;
11. No swallowing difficulties; No shoulder joint movement disorders;
12. Complete clinical data.

Exclusion Criteria:

1. Age<16 years old, still in puberty, or disease duration ≤ 1 year;
2. Simple obesity, no obvious glandular tissue was found on breast ultrasound examination;
3. Male patients with breast developmental disorders secondary to other diseases;
4. Patients with contraindications for general anesthesia surgery such as coagulation dysfunction and severe cardiovascular disease, who cannot tolerate surgery;
5. The clinical data is basically incomplete;
6. Other surgical methods;
7. Individuals with a history of breast surgery or breast tumors in the past;
8. The serious diseases of non malignant tumors such as congenital testicular hypoplasia syndrome, cirrhosis, primary hypogonadism, and hyperthyroidism will affect the patient's compliance or put the patient in a dangerous state;
9. Dementia, intellectual disability, or any mental illness that hinders understanding of informed consent forms;
10. Lack of trust in surgical outcomes and weak desire for surgery.

Ages: 17 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Patient's and doctor's satisfaction | 2 years
  Use the Health Status Survey Questionnaire (SF-36) to assess the general condition of patients.
Patient's psychological status using the Self Rating Anxiety Scale (SAS) | 2 years
  Use the Self Rating Anxiety Scale (SAS) to assess the psychological status of patients.
Patient's psychological status | 2 years
  Use the Self Rating Depression Scale (SDS) to assess the psychological status of patients.
Patient's sensory | 2 years
  Using Semmes Weinstein (S-W) monofilament to detect postoperative sensory recovery in patients.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol